CLINICAL TRIAL: NCT04840888
Title: Evaluation of the Effect of Food, Omeprazole, Itraconazole, and Carbamazepine on the Pharmacokinetics of LY3484356 in Healthy Females of Non-Child-Bearing Potential
Brief Title: A Study of LY3484356 in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18204; J2J-MC-JZLD (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Imlunestrant; Omeprazole; Itraconazole; Carbamazepine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 Sequence 1: 400 mg LY3484356 Fasted/ 400 mg LY3484356 Fed (Experimental): Participants were randomized (1:1) to 1 of 2 treatment sequences; LY3484356 administered as single doses orally with (fed) or without food (fasted) as below:
  Period 1: Single dose of 400 mg LY3484356 in the fasted state. Period 2: Single dose of 400 mg LY3484356 in the fed state. There was a washout period of 4 days between doses of LY3484356
  Interventions: Drug: LY3484356
- Cohort 1 Sequence 2: 400 mg LY3484356 Fed/ 400 mg LY3484356 Fasted (Experimental): Participants were randomized (1:1) to 1 of 2 treatment sequences; LY3484356 administered as single doses orally with (fed) or without food (fasted) as below:
  Period 1: Single dose of 400 mg LY3484356 in the fed state. Period 2: Single dose of 400 mg LY3484356 in the fasted state. There was a washout period of 4 days between doses of LY3484356.
  Interventions: Drug: LY3484356
- Cohort 2: LY3484356 + Omeprazole (Experimental): Participants received single dose of LY3484356 and a single dose of omeprazole alone and in combination administered orally as below:
  Day 1: 400 mg LY3484356 alone Days 5 to 8: 40 mg omeprazole alone once daily Day 9: 400 mg LY3484356 + 40 mg omeprazole once There was a washout period of 8 days between doses of LY3484356.
  Interventions: Drug: LY3484356; Drug: Omeprazole
- Cohort 3: LY3484356 + Itraconazole (Experimental): Participants received single dose of LY3484356 and a single dose of Itraconazole alone and in combination administered orally as below:
  Day 1: 200 mg LY3484356 alone Days 5 to 9: 200 mg itraconazole alone (twice on Day 5 [dose separated by approximately 12 hours], then once daily on Days 6 through 9) Day 10: 200 mg LY3484356 + 200 mg itraconazole once (coadministered with the morning dose) Days 11 to 16: 200 mg itraconazole alone once daily. There was a washout period of 9 days between doses of LY3484356.
  Interventions: Drug: LY3484356; Drug: Itraconazole
- Cohort 4: LY3484356 + Carbamazepine (Experimental): Participants received single dose of LY3484356 and a single dose of carbamazepine alone and in combination administered orally as below:
  Day 1: 400 mg LY3484356 alone Days 6 to 8: 100 mg carbamazepine BID alone Days 9 to 11: 200 mg carbamazepine BID alone Days 12 to 17: 300 mg carbamazepine BID alone Day 18: 300 mg carbamazepine BID + 400 mg LY3484356 (coadministered with morning dose) Days 19 to 22: 300 mg carbamazepine BID alone Day 23: 300 mg carbamazepine alone (morning dose only). There was a washout period of 17 days between doses of LY3484356.
  Interventions: Drug: LY3484356; Drug: Carbamazepine
- Cohort 5: Carbamazepine + Midazolam (Experimental): Participants received single dose of Carbamazepine and a single dose of midazolam alone and in combination administered orally as below:
  Day 1: 1.2 mg midazolam alone Days 2 to 4: 100 mg carbamazepine BID alone Days 5 to 7: 200 mg carbamazepine BID alone Days 8 to 10: 300 mg carbamazepine BID alone Day 11: 300 mg carbamazepine BID + 1.2 mg midazolam (coadministered with morning dose) Days 12 to 13: 300 mg carbamazepine BID alone Day 14: 300 mg carbamazepine BID + 1.2 mg midazolam (coadministered with morning dose).
  Interventions: Drug: Carbamazepine; Drug: Midazolam

INTERVENTIONS:
Drug: LY3484356 — Administered orally.
  Arms: Cohort 1 Sequence 1: 400 mg LY3484356 Fasted/ 400 mg LY3484356 Fed; Cohort 1 Sequence 2: 400 mg LY3484356 Fed/ 400 mg LY3484356 Fasted; Cohort 2: LY3484356 + Omeprazole; Cohort 3: LY3484356 + Itraconazole; Cohort 4: LY3484356 + Carbamazepine
Drug: Omeprazole — Administered orally.
  Arms: Cohort 2: LY3484356 + Omeprazole
Drug: Itraconazole — Administered orally.
  Arms: Cohort 3: LY3484356 + Itraconazole
Drug: Carbamazepine — Administered orally.
  Arms: Cohort 4: LY3484356 + Carbamazepine; Cohort 5: Carbamazepine + Midazolam
Drug: Midazolam — Administered orally.
  Arms: Cohort 5: Carbamazepine + Midazolam

SUMMARY:
The main purpose of this study is to evaluate the amount of LY3484356 that is found in the blood stream and how long the body takes to get rid of it when given with and without food. Participants are healthy females of non-childbearing potential. The study will also evaluate the tolerability and safety of LY3484356 by collecting the information about any side effects that may occur. The participant's involvement with the study will last approximately 27 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical assessment
* Body mass index (BMI) within the range 18.0 to 35.0 kilograms per meter squared (kg/m²)
* Female participants of non childbearing potential. This includes females who are not pregnant, non-lactating and either: Infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy or bilateral salpingectomy, bilateral tubal ligation, or bilateral tubal occlusion), or alternate medical cause/congenital anomaly (for example, Müllerian agenesis) or postmenopausal

Exclusion Criteria:

* Have a history or presence of cardiovascular (eg, symptomatic bradycardia with resting heart rate of <60 beats per minute), respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Show evidence of hepatitis B, evidence of hepatitis C and/or have evidence of human immunodeficiency virus (HIV) infection
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing
* Use or intend to use medications that inhibit or induce CYP3A4 within 14 days prior to dosing until completion of the follow-up visit
* Smoke more than 10 cigarettes or use the equivalent tobacco, smoking-cessation products, nicotine-containing products, or e cigarettes (nicotine and non nicotine) per day

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - Covance Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Sequence 1: 400 mg LY3484356 Fasted/ 400 mg LY3484356 Fed: Participants were randomized (1:1) to 1 of 2 treatment sequences; LY3484356 received as single dose with (fed) or without food (fasted) administered orally as below:
  Period 1: Single dose of 400 mg LY3484356 in the fasted state.
  Period 2: Single dose of 400 mg LY3484356 in the fed state.
  There was a washout period of 4 days between doses of LY3484356
- Cohort 1 Sequence 2: 400 mg LY3484356 Fed/ 400 mg LY3484356 Fasted: Participants were randomized (1:1) to 1 of 2 treatment sequences; LY3484356 received as single dose with (fed) or without food (fasted) administered orally as below:
  Period 1: Single dose of 400 mg LY3484356 in the fed state.
  Period 2: Single dose of 400 mg LY3484356 in the fasted state.
  There was a washout period of 4 days between doses of LY3484356.
- Cohort 2: LY3484356 + Omeprazole: Participants received single dose of LY3484356 and a single oral dose of omeprazole alone and in combination administered orally as below:
  Day 1: 400 mg LY3484356 alone
  Days 5 to 8: 40 mg omeprazole alone once daily
  Day 9: 400 mg LY3484356 + 40 mg omeprazole once
  There was a washout period of 8 days between doses of LY3484356.
- Cohort 3: LY3484356 + Itraconazole: Participants received single dose of LY3484356 and a single oral dose of Itraconazole alone and in combination administered orally as below:
  Day 1: 200 mg LY3484356 alone
  Days 5 to 9: 200 mg itraconazole alone (twice on Day 5 [dose separated by approximately 12 hours], then once daily on Days 6 through 9)
  Day 10: 200 mg LY3484356 + 200 mg itraconazole once (coadministered with the morning dose)
  Days 11 to 16: 200 mg itraconazole alone once daily.
  There was a washout period of 9 days between doses of LY3484356.
- Cohort 4: LY3484356 + Carbamazepine: Participants received single dose of LY3484356 and a single oral dose of carbamazepine alone and in combination administered orally as below:
  Day 1: 400 mg LY3484356 alone
  Days 6 to 8: 100 mg carbamazepine twice daily (BID) alone
  Days 9 to 11: 200 mg carbamazepine BID alone
  Days 12 to 17: 300 mg carbamazepine BID alone
  Day 18: 300 mg carbamazepine BID + 400 mg LY3484356 (coadministered with morning dose)
  Days 19 to 22: 300 mg carbamazepine BID alone
  Day 23: 300 mg carbamazepine alone (morning dose only).
  There was a washout period of 17 days between doses of LY3484356.
- Cohort 5: Carbamazepine + Midazolam: Participants received single dose of Carbamazepine and a single oral dose of midazolam alone and in combination administered orally as below:
  Day 1: 1.2 mg midazolam alone
  Days 2 to 4: 100 mg carbamazepine BID alone
  Days 5 to 7: 200 mg carbamazepine BID alone
  Days 8 to 10: 300 mg carbamazepine BID alone
  Day 11: 300 mg carbamazepine BID + 1.2 mg midazolam (coadministered with morning dose)
  Days 12 to 13: 300 mg carbamazepine BID alone
  Day 14: 300 mg carbamazepine BID + 1.2 mg midazolam (coadministered with morning dose).
Period: Period 1
Arm/Group | Cohort 1 Sequence 1: 400 mg LY3484356 Fasted/ 400 mg LY3484356 Fed | Cohort 1 Sequence 2: 400 mg LY3484356 Fed/ 400 mg LY3484356 Fasted | Cohort 2: LY3484356 + Omeprazole | Cohort 3: LY3484356 + Itraconazole | Cohort 4: LY3484356 + Carbamazepine | Cohort 5: Carbamazepine + Midazolam
Started | 5 | 3 | 10 | 20 | 29 | 15
Received at Least One Dose of Study Drug | 5 | 3 | 10 | 20 | 29 | 15
Completed | 5 | 3 | 9 | 19 | 18 | 14
Not Completed | 0 | 0 | 1 | 1 | 11 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 10 | 1
Period: Period 2
Arm/Group | Cohort 1 Sequence 1: 400 mg LY3484356 Fasted/ 400 mg LY3484356 Fed | Cohort 1 Sequence 2: 400 mg LY3484356 Fed/ 400 mg LY3484356 Fasted | Cohort 2: LY3484356 + Omeprazole | Cohort 3: LY3484356 + Itraconazole | Cohort 4: LY3484356 + Carbamazepine | Cohort 5: Carbamazepine + Midazolam
Started | 5 | 3 | 0 (Per analysis, Cohort 2 participants were assigned only to treatment period 1.) | 0 (Per analysis, Cohort 3 participants were assigned only to treatment period 1.) | 0 (Per analysis, Cohort 4 participants were assigned only to treatment period 1.) | 0 (Per analysis, Cohort 5 participants were assigned only to treatment period 1.)
Received at Least One Dose of Study Drug | 5 | 3 | 0 | 0 | 0 | 0
Completed | 5 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Cohort 1: Sequence 1/Sequence 2: Participants were randomized (1:1) to 1 of 2 treatment sequences; LY3484356 received as single dose with (fed) or without food (fasted) administered orally as below:
  Cohort 1 Sequence 1:
  Period 1: Single dose of 400 mg LY3484356 in the fed state.
  Period 2: Single dose of 400 mg LY3484356 in the fasted state.
  Cohort 1 Sequence 2:
  Period 1: Single dose of 400 mg LY3484356 in the fasted state.
  Period 2: Single dose of 400 mg LY3484356 in the fed state.
  There was a washout period of 4 days between doses of LY3484356
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Sequence 1/Sequence 2 | Cohort 2: LY3484356 + Omeprazole | Cohort 3: LY3484356 + Itraconazole | Cohort 4: LY3484356 + Carbamazepine | Cohort 5: Carbamazepine + Midazolam | Total
Number analyzed (Participants) | 8 | 10 | 20 | 29 | 15 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (6.9) | 58.6 (6.9) | 52.5 (9.2) | 49.8 (10.1) | 46.4 (10.4) | 51.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 20 | 29 | 3 | 70
  Male | 0 | 0 | 0 | 0 | 12 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 11 | 18 | 8 | 45
  Not Hispanic or Latino | 5 | 5 | 9 | 11 | 7 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 8 | 2 | 18
  White | 4 | 7 | 18 | 21 | 13 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 20 | 29 | 15 | 82

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3484356 (Cohort 1)
Description: PK: AUC[0-∞] of LY3484356
Time Frame: Period 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours (h) postdose; Period 2: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 and 96 h postdose
Population: All enrolled participants in cohort 1 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Cohort 1: 400 mg LY3484356 Fasted: Participants received single oral dose of 400 mg LY3484356 in the fasted state.
- Cohort 1: 400 mg LY3484356 Fed: Participants received single oral dose of 400 mg LY3484356 in the fed state.
Arm/Group | Cohort 1: 400 mg LY3484356 Fasted | Cohort 1: 400 mg LY3484356 Fed
Number analyzed (Participants) | 4 | 6
nanogram*hour per milliliter (ng*hr/mL) | 1810 (59) | 4350 (39)

2. Primary Outcome: PK: AUC[0-∞] of LY3484356 (Cohort 2)
Description: PK: AUC[0-∞] of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 9: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 2 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 2: LY3484356 + Omeprazole
Number analyzed (Participants) | 4
ng*hr/mL
  Day 1 | 2270 (93)
  Day 9 | 1960 (46)

3. Primary Outcome: PK: AUC[0-∞] of LY3484356 (Cohort 3)
Description: PK: AUC[0-∞] of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 10: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 3 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 3: LY3484356 + Itraconazole
Number analyzed (Participants) | 19
ng*hr/mL
  Day 1: number analyzed (Participants) | 14
  Day 1 | 1430 (58)
  Day 10 | 3120 (41)

4. Primary Outcome: PK: AUC[0-∞] of LY3484356 (Cohort 4)
Description: AUC[0-∞] of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 18: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 4 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 4: LY3484356 + Carbamazepine
Number analyzed (Participants) | 26
ng*hr/mL
  Day 1 | 1950 (67)
  Day 18: number analyzed (Participants) | 24
  Day 18 | 1090 (32)

5. Primary Outcome: PK: Time of Maximum Observed Concentration (Tmax) of LY3484356 (Cohort 1)
Description: PK: Tmax of LY3484356
Time Frame: Period 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 h postdose; Period 2: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 and 96 h postdose
Population: All enrolled participants in cohort 1 who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: 400 mg LY3484356 Fasted | Cohort 1: 400 mg LY3484356 Fed
Number analyzed (Participants) | 8 | 8
hours | 8.00 [3.00 to 35.80] | 3.02 [2.00 to 8.00]

6. Primary Outcome: PK: Tmax of LY3484356 (Cohort 2)
Description: PK: Tmax of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 9: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 2 who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 2: LY3484356 + Omeprazole
Number analyzed (Participants) | 10
hours
  Day 1 | 6.02 [1.00 to 10.00]
  Day 9: number analyzed (Participants) | 9
  Day 9 | 6.00 [4.00 to 36.00]

7. Primary Outcome: PK: Tmax of LY3484356 (Cohort 3)
Description: PK: Tmax of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 10: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 3 who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 3: LY3484356 + Itraconazole
Number analyzed (Participants) | 20
hours
  Day 1 | 6.00 [2.00 to 36.00]
  Day 10 | 6.00 [1.00 to 12.00]

8. Primary Outcome: PK: Tmax of LY3484356 (Cohort 4)
Description: Tmax of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 18: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 4 who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 4: LY3484356 + Carbamazepine
Number analyzed (Participants) | 29
hours
  Day 1 | 4.00 [2.00 to 36.00]
  Day 18: number analyzed (Participants) | 25
  Day 18 | 3.87 [1.00 to 8.00]

9. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of LY3484356 (Cohort 1)
Description: Cmax of LY3484356
Time Frame: as for outcome 5
Population: All enrolled participants in cohort 1 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | Cohort 1: 400 mg LY3484356 Fasted | Cohort 1: 400 mg LY3484356 Fed
Number analyzed (Participants) | 8 | 8
nanogram per millilitre (ng/mL) | 37.2 (51) | 143 (28)

10. Primary Outcome: PK: Cmax of LY3484356 (Cohort 2)
Description: Cmax of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 9: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 2 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 2: LY3484356 + Omeprazole
Number analyzed (Participants) | 10
ng/mL
  Day 1 | 49.1 (61)
  Day 9: number analyzed (Participants) | 9
  Day 9 | 39.6 (47)

11. Primary Outcome: PK: Cmax of LY3484356 (Cohort 3)
Description: Cmax of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 10: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 3 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 3: LY3484356 + Itraconazole: Participants received single dose of LY3484356 and a single dose of Itraconazole alone and in combination administered orally as below:
  Day 1: 200 mg LY3484356 alone
  Days 5 to 9: 200 mg itraconazole alone (twice on Day 5 [dose separated by approximately 12 hours], then once daily on Days 6 through 9)
  Day 10: 200 mg LY3484356 + 200 mg itraconazole once (coadministered with the morning dose).
  Days 11 to 16: 200 mg itraconazole alone once daily.
  There was a washout period of 9 days between doses of LY3484356.
Arm/Group | Cohort 3: LY3484356 + Itraconazole
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 30.3 (57)
  Day 10 | 56.7 (47)

12. Primary Outcome: PK: Cmax of LY3484356 (Cohort 4)
Description: Cmax of LY3484356
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose; Day 18: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 h postdose
Population: All enrolled participants in cohort 4 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 4: LY3484356 + Carbamazepine
Number analyzed (Participants) | 29
ng/mL
  Day 1 | 49.6 (76)
  Day 18: number analyzed (Participants) | 25
  Day 18 | 33.3 (41)

ADVERSE EVENTS:
Time Frame: Cohort 1: up to 19 days, Cohort 2: up to 24 days, Cohort 3: up to 27 days, Cohort 4: up to 37 days, and Cohort 5: up to 25 days
Description: All enrolled participants who received at least one dose of study drug. Based on the planned safety analysis, adverse events were collected per each dose level of treatment regimen
Groups:
- Cohort 2: 400 mg LY3484356 (Day 1): Participants received 400 mg LY3484356 alone administered orally (Day 1).
- Cohort 2: 40 mg Omeprazole (Days 5 to 8): Participants received 40 mg omeprazole administered orally once daily (Days 5 to 8).
- Cohort 2: 400 mg LY3484356 + 40 mg Omeprazole (Day 9): Participants received 400 mg LY3484356 + 40 mg omeprazole administered orally (Day 9).
- Cohort 3: 200 mg LY3484356 (Day 1): Participants received 200 mg LY3484356 administered orally (Day 1)
- Cohort 3: 200 mg Itraconazole (Days 5 to 9): Participants received 200 mg itraconazole administered orally alone (twice on Day 5 [dose separated by approximately 12 hours], then once daily on Days 6 through 9)
- Cohort 3: 200 mg LY3484356 + 200 mg Itraconazole (Days 10 to 16): Participants received 200 mg LY3484356 + 200 mg itraconazole administered orally once (co-administered with the morning dose) (Day 10), then 200 mg itraconazole administered orally alone once daily (Days 11 to 16).
- Cohort 4: 400 mg LY3484356 (Day 1): Participants received 400 mg LY3484356 administered orally (Day 1)
- Cohort 4: 100 mg Carbamazepine (Days 6 to 8): Participants received 100 mg carbamazepine administered orally BID (Days 6 to 8).
- Cohort 4: 200 mg Carbamazepine (Days 9 to 11): Participants received 200 mg carbamazepine administered orally BID (Days 9 to 11).
- Cohort 4: 300 mg Carbamazepine + 400 mg LY3484356 (Days 12 to 22): Participants received 300 mg carbamazepine administered orally BID (Days 12 to 17), then 300 mg carbamazepine BID + 400 mg LY3484356 (co-administered with morning dose) administered orally (Day 18) followed by 300 mg carbamazepine administered orally BID (Day 19 to 22).
- Cohort 4: 300 mg Carbamazepine (Day 23): Participants received 300 mg carbamazepine (morning dose only) administered orally (Day 23).
- Cohort 5: 1.2 mg Midazolam (Day 1): Participants received 1.2 mg midazolam administered orally (Day 1).
- Cohort 5: 100 mg Carbamazepine (Days 2 to 4): Participants received 100 mg carbamazepine administered orally BID (Days 2 to 4).
- Cohort 5: 200 mg Carbamazepine (Days 5 to 7): Participants received 200 mg carbamazepine administered orally BID (Days 5 to 7).
- Cohort 5: 300 mg Carbamazepine (Days 8 to 10): Participants received 300 mg carbamazepine administered orally BID (Days 8 to 10).
- Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 11): Participants received 300 mg carbamazepine BID + 1.2 mg midazolam (co-administered with morning dose) administered orally (Day 11)
- Cohort 5: 300 mg Carbamazepine (Days 12 to 13): Participants received 300 mg carbamazepine administered orally BID (Days 12 to 13)
- Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 14): Participants received 300 mg carbamazepine BID + 1.2 mg midazolam (co-administered with morning dose) administered orally (Day 14).
Arm/Group | Cohort 1: 400 mg LY3484356 Fasted | Cohort 1: 400 mg LY3484356 Fed | Cohort 2: 400 mg LY3484356 (Day 1) | Cohort 2: 40 mg Omeprazole (Days 5 to 8) | Cohort 2: 400 mg LY3484356 + 40 mg Omeprazole (Day 9) | Cohort 3: 200 mg LY3484356 (Day 1) | Cohort 3: 200 mg Itraconazole (Days 5 to 9) | Cohort 3: 200 mg LY3484356 + 200 mg Itraconazole (Days 10 to 16) | Cohort 4: 400 mg LY3484356 (Day 1) | Cohort 4: 100 mg Carbamazepine (Days 6 to 8) | Cohort 4: 200 mg Carbamazepine (Days 9 to 11) | Cohort 4: 300 mg Carbamazepine + 400 mg LY3484356 (Days 12 to 22) | Cohort 4: 300 mg Carbamazepine (Day 23) | Cohort 5: 1.2 mg Midazolam (Day 1) | Cohort 5: 100 mg Carbamazepine (Days 2 to 4) | Cohort 5: 200 mg Carbamazepine (Days 5 to 7) | Cohort 5: 300 mg Carbamazepine (Days 8 to 10) | Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 11) | Cohort 5: 300 mg Carbamazepine (Days 12 to 13) | Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 14)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/9 | 0/20 | 0/20 | 0/20 | 0/29 | 0/28 | 0/28 | 0/28 | 0/20 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/9 | 0/20 | 0/20 | 0/20 | 0/29 | 0/28 | 0/28 | 1/28 | 0/20 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 2/10 | 2/10 | 1/9 | 5/20 | 8/20 | 2/20 | 2/29 | 1/28 | 6/28 | 16/28 | 3/20 | 0/15 | 1/15 | 0/15 | 2/15 | 1/15 | 2/15 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 400 mg LY3484356 Fasted (N=8) | Cohort 1: 400 mg LY3484356 Fed (N=8) | Cohort 2: 400 mg LY3484356 (Day 1) (N=10) | Cohort 2: 40 mg Omeprazole (Days 5 to 8) (N=10) | Cohort 2: 400 mg LY3484356 + 40 mg Omeprazole (Day 9) (N=9) | Cohort 3: 200 mg LY3484356 (Day 1) (N=20) | Cohort 3: 200 mg Itraconazole (Days 5 to 9) (N=20) | Cohort 3: 200 mg LY3484356 + 200 mg Itraconazole (Days 10 to 16) (N=20) | Cohort 4: 400 mg LY3484356 (Day 1) (N=29) | Cohort 4: 100 mg Carbamazepine (Days 6 to 8) (N=28) | Cohort 4: 200 mg Carbamazepine (Days 9 to 11) (N=28) | Cohort 4: 300 mg Carbamazepine + 400 mg LY3484356 (Days 12 to 22) (N=28) | Cohort 4: 300 mg Carbamazepine (Day 23) (N=20) | Cohort 5: 1.2 mg Midazolam (Day 1) (N=15) | Cohort 5: 100 mg Carbamazepine (Days 2 to 4) (N=15) | Cohort 5: 200 mg Carbamazepine (Days 5 to 7) (N=15) | Cohort 5: 300 mg Carbamazepine (Days 8 to 10) (N=15) | Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 11) (N=15) | Cohort 5: 300 mg Carbamazepine (Days 12 to 13) (N=15) | Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 14) (N=14)
Hepatitis e (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 400 mg LY3484356 Fasted (N=8) | Cohort 1: 400 mg LY3484356 Fed (N=8) | Cohort 2: 400 mg LY3484356 (Day 1) (N=10) | Cohort 2: 40 mg Omeprazole (Days 5 to 8) (N=10) | Cohort 2: 400 mg LY3484356 + 40 mg Omeprazole (Day 9) (N=9) | Cohort 3: 200 mg LY3484356 (Day 1) (N=20) | Cohort 3: 200 mg Itraconazole (Days 5 to 9) (N=20) | Cohort 3: 200 mg LY3484356 + 200 mg Itraconazole (Days 10 to 16) (N=20) | Cohort 4: 400 mg LY3484356 (Day 1) (N=29) | Cohort 4: 100 mg Carbamazepine (Days 6 to 8) (N=28) | Cohort 4: 200 mg Carbamazepine (Days 9 to 11) (N=28) | Cohort 4: 300 mg Carbamazepine + 400 mg LY3484356 (Days 12 to 22) (N=28) | Cohort 4: 300 mg Carbamazepine (Day 23) (N=20) | Cohort 5: 1.2 mg Midazolam (Day 1) (N=15) | Cohort 5: 100 mg Carbamazepine (Days 2 to 4) (N=15) | Cohort 5: 200 mg Carbamazepine (Days 5 to 7) (N=15) | Cohort 5: 300 mg Carbamazepine (Days 8 to 10) (N=15) | Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 11) (N=15) | Cohort 5: 300 mg Carbamazepine (Days 12 to 13) (N=15) | Cohort 5: 300 mg Carbamazepine + 1.2 mg Midazolam (Day 14) (N=14)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04840888/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT04840888/SAP_001.pdf